CLINICAL TRIAL: NCT06594393
Title: A Randomized, Double-blind, Vehicle-controlled Phase 2 Study to Evaluate Efficacy, Safety, and Tolerability of Topically Applied TCP-25 in Patients With Epidermolysis Bullosa
Brief Title: A Phase 2 Study of TCP-25 Gel in Patients With Epidermolysis Bullosa, STEP-study
Acronym: STEP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xinnate AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCP25-002
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Epidermolysis Bullosa (EB); Dystrophic Epidermolysis Bullosa; Junctional Epidermolysis Bullosa
Keywords: epidermolysis bullosa; topical treatment
MeSH Terms: conditions — Epidermolysis Bullosa; Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa, Junctional

STUDY DESIGN:
Intervention Model Description: Intra-subject control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCP-25 (Experimental): Topical gel
  Interventions: Drug: TCP-25 gel
- Vehicle (Placebo Comparator): Placebo gel
  Interventions: Drug: Vehicle (placebo)

INTERVENTIONS:
Drug: TCP-25 gel — Topical gel
  Arms: TCP-25
Drug: Vehicle (placebo) — Placebo gel
  Arms: Vehicle

SUMMARY:
This is a Phase 2, double-blind, randomized, vehicle-controlled study designed to evaluate efficacy, safety, and tolerability of topically applied TCP-25 gel in patients with confirmed DEB or JEB. The study will implement intrasubject randomization, ie, a pair of matching index wounds will be randomly assigned to be treated with a local application of either TCP 25 gel or vehicle gel.

DETAILED DESCRIPTION:
The study will include a Screening Period, a Treatment Period (Days 1 to 56, with study visits conducted every 2 weeks, including the baseline [Day 1], Day 14, Day 28, Day 42, and Day 56 visits) and a Safety Follow-up conducted via a telephone/video call at approximately 14 days after the last dose of the IMP. Patients will undergo efficacy, safety, tolerability, and PK assessments at scheduled visits. For evaluation of the primary efficacy endpoint, a trained clinician will take the images of the index wounds at all scheduled visits from baseline through Day 56 (Visit 6) using 3D digital photography and software for wound measurement.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with documented diagnosis of DEB or JEB, confirmed by genetic testing and/or by a skin biopsy with immunofluorescence mapping.
* Patients ≥4 years old. Note: Initially, patients ≥12 years will be enrolled. Enrollment will be open to 4 to 11 year old pediatric patients (both inclusive), after a DMC reviews and provides a positive opinion regarding the safety and tolerability of the IMP in at least 3 patients 12 to 18 years old who have completed at least 4 weeks of IMP use.

Exclusion Criteria:

* The patient has any subtype of EB other than DEB or JEB.
* The patient is currently being treated or planned to be treated with systemic antibiotics.

Note: Use of preventive and/or anti-inflammatory antibiotic treatment, including doxycycline, on an established treatment regimen (stable dose for ≥6 weeks before the Baseline Visit) is permitted. Use of topical antibiotics on the index wounds within 7 days before the Baseline Visit is prohibited.

• Use of systemic corticosteroids >0.2 mg/kg prednisone dose equivalent per day within 30 days or use of topical corticosteroids on index wounds within 7 days before the Screening Visit.

Note: Corticosteroids for inhalation, ophthalmic, or intranasal use are permitted.

• The patient has a history of or current malignancy over the index wound, eg, basal cell carcinoma or squamous cell carcinoma.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Open wound area | 56 days

SECONDARY OUTCOMES:
Frequency, intensity, and seriousness of Adverse Events in all treated patients until end of treatment | 56 days
Change in procedural pain using the Wong Baker FACES® Pain Rating Scale (0 min -10 max) | 56 days
  Wong Baker FACES pain rating scale uses 6 graphically or cartoon-depicted faces with varying facial expressions that represent no pain (no hurt) (Face 0) to worst pain/hurt that can be imagined (Face 10).
Change from baseline in clinical impression of overall treatment area | 56 days
TCP-25 plasma concentrations | 56 days
Number of participants with treatment-related local tolerability assessment at the area of IMP application assessed on a 4-point scale | 56 days
Clinically significant changes from baseline in blood pressure until end of treatment | 56 days
Number of patients with clinically significant changes from baseline in pulse rate until end of treatment | 56 days
Number of patients with clinically significant changes from baseline in physical examination findings until end of treatment | 56 days

CONTACTS AND LOCATIONS:
Locations (6):
- Hopital St Louis, Paris, France
- Greece (2):
  - Andreas Syngros Hospital of Veneral & Dermatological Diseases, Athens
  - Hospital Of Skin And Venereal Diseases of Thessaloniki, Thessaloniki
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Univ La Paz, Madrid
- University hospital, Lund, Skåne County, Sweden

REFERENCES:
- [Background] Lundgren S, Wallblom K, Fisher J, Erdmann S, Schmidtchen A, Saleh K. Study protocol for a phase 1, randomised, double-blind, placebo-controlled study to investigate the safety, tolerability and pharmacokinetics of ascending topical doses of TCP-25 applied to epidermal suction blister wounds in healthy male and female volunteers. BMJ Open. 2023 Feb 22;13(2):e064866. doi: 10.1136/bmjopen-2022-064866. PMID 36813496